CLINICAL TRIAL: NCT05048719
Title: A Phase 2 Study of Once-Daily LY3502970 Compared With Placebo and Once-Weekly Dulaglutide in Participants With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3502970 in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17787; J2A-MC-GZGE (Other: Eli Lilly and Company); 2021-002806-29 (EudraCT Number)
Record Dates: First submitted 2021-09-13; First posted 2021-09-17 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — orforglipron; dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- 3 milligrams (mg) LY3502970 (Experimental): Participants received maintenance dose of 3 mg with dose escalation starting from 2 mg LY3502970 administered orally once daily (QD).
  Interventions: Drug: LY3502970
- 12 mg LY3502970 (Experimental): Participants received maintenance dose 12 mg with dose escalation starting from 2 mg, 6 mg and then 12 mg LY3502970 administered orally QD.
  Interventions: Drug: LY3502970
- 24 mg LY3502970 (Experimental): Participants received maintenance dose 24 mg with dose escalation starting from 3 mg, 6 mg, 8 mg,12 mg and then 24 mg LY3502970 administered orally QD.
  Interventions: Drug: LY3502970
- 36 mg LY3502970 - 1 (Experimental): Participants received maintenance dose 36 mg with dose escalation starting from 2 mg, 3 mg, 6 mg, 8 mg, 12 mg, 24 mg and then 36 mg LY3502970 administered orally QD.
  Interventions: Drug: LY3502970
- 36 mg LY3502970 - 2 (Experimental): Participants received maintenance dose 36 mg with dose escalation starting from 3 mg, 6 mg,12 mg, 24 mg and then 36 mg LY3502970 administered orally QD.
  Interventions: Drug: LY3502970
- 45 mg LY3502970 - 1 (Experimental): Participants received maintenance dose 45 mg with dose escalation starting from 3 mg, 6 mg, 8 mg, 12 mg, 24 mg, 36 mg and then 45 mg LY3502970 administered orally QD.
  Interventions: Drug: LY3502970
- 45 mg LY3502970 - 2 (Experimental): Participants received maintenance dose 45 mg with dose escalation starting from 2 mg, 3 mg, 6 mg, 12 mg, 24 mg, 36 mg and then 45 mg LY3502970 administered orally QD.
  Interventions: Drug: LY3502970
- 1.5 mg Dulaglutide (Active Comparator): Participants received 1.5 mg Dulaglutide administered subcutaneously (SC) once weekly (QW).
  Interventions: Drug: Dulaglutide
- Placebo (Placebo Comparator): Participants received matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3502970 — Administered orally
  Arms: 12 mg LY3502970; 24 mg LY3502970; 3 milligrams (mg) LY3502970; 36 mg LY3502970 - 1; 36 mg LY3502970 - 2; 45 mg LY3502970 - 1; 45 mg LY3502970 - 2
Drug: Dulaglutide — Administered subcutaneously
  Arms: 1.5 mg Dulaglutide
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Placebo — Administered subcutaneously
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of LY3502970 in participants with type 2 diabetes (T2D) who failed to achieve adequate glycemic control on diet and exercise alone or on a stable dose of metformin. This study will last about 30 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with Type 2 Diabetes on diet and exercise and/or a stable dose of metformin
* Have a stable body weight for the 3 months prior to randomization
* Have a body mass index (BMI) ≥23 kilogram/square meter (kg/m²)
* Males must agree to use highly effective methods of contraception
* Women not of childbearing potential (WNOCBP) may participate in this trial
* Note: Hormone replacement therapy in post-menopausal women is allowed but women must be on stable therapy for 3 months prior to day 1.

Exclusion Criteria:

* Have Type 1 diabetes mellitus (T1DM) or history of ketoacidosis or hyperosmolar coma
* Have a history of diabetic retinopathy, diabetic maculopathy, or severe non-proliferative diabetic retinopathy that requires immediate treatment intervention
* Have had more than 1 episode of severe hypoglycemia and aware of hypoglycemic symptoms
* Have acute or chronic pancreatitis
* Have obesity induced other endocrine disorders (Cushing's syndrome or Prader - Willi syndrome)
* Have gastric emptying abnormality or chronically take medications impacting GI motility
* Have poorly controlled hypertension
* Have the following heart conditions within the last 6 months: myocardial infarction (MI), unstable angina, coronary artery bypass graft, percutaneous coronary intervention (diagnostic angiograms are permitted), transient ischemic attack (TIA), cerebrovascular accident (stroke)or decompensated congestive heart failure, or IV heart failure
* Have any symptoms of other liver diseases besides nonalcoholic fatty liver disease (NAFLD)
* Have HIV, or Hepatitis B or Hepatitis C

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (44):
- United States (20):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research, Westlake, Los Angeles, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - Touro University California, Vallejo, California
  - New West Physicians Clinical Research, Golden, Colorado
  - Optumcare Colorado Springs - Monument, Monument, Colorado
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Clinvest Research LLC, Springfield, Missouri
  - Premier Research, Trenton, New Jersey
  - Intend Research, LLC, Norman, Oklahoma
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Family Medical Associates, Levittown, Pennsylvania
  - Tristar Clinical Investigations, Philadelphia, Pennsylvania
  - Dallas Diabetes Research Center, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Bandera Family Health Care, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Capital Clinical Research Center, Olympia, Washington
  - Eastside Research Associates, Redmond, Washington
- Hungary (8):
  - Bugát Pál Kórház, Gyöngyös, Heves County
  - Kanizsai Dorottya Korhaz, Nagykanizsa, Zala County
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg, Zala County
  - Szent Margit Rendelőintézet Nonprofit Kft, Budapest
  - Clinexpert Kft., Budapest
  - ClinDiab Kft., Budapest
  - TRANTOR'99 Bt. Anyagcsere Centrum, Budapest
  - Strazsahegy Medicina Bt., Budapest
- Poland (8):
  - Centrum Zdrowia Tuchów, Wierzchosławice, Lesser Poland Voivodeship
  - Wojewódzki Zespól Specjalistycznej Opieki Zdrowotnej, Wroclaw, Lower Silesian Voivodeship
  - Gabinety TERPA, Lublin, Lublin Voivodeship
  - NZOZ Medica, Lublin, Lublin Voivodeship
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw, Masovian Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - NZOZ Przychodnia Specjalistyczna Andrzej Wittek, Henryk Rudzki, Ruda Śląska, Silesian Voivodeship
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz, Łódź Voivodeship
- Puerto Rico (3):
  - Dorado Medical Complex, Dorado
  - Clinical Research Management Group Inc. - Hospital San Cristobal, Ponce
  - BRCR Global Puerto Rico-Unda, San Juan
- Slovakia (5):
  - Ambulancia diabetológie a porúch látkovej premeny a výživy - DIABEDA, Bratislava, Bratislava Region
  - Diabetol, Prešov, Presov
  - MEDI-DIA s.r.o., Sabinov, Presov
  - DIA-MED CENTRUM s.r.o., Púchov, Trenčín Region
  - Funkystuff, Nové Zámky

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Wharton S, Rosenstock J, Konige M, Lin Y, Duffin K, Wilson J, Banerjee H, Pirro V, Kazda C, Mather K. Treatment with orforglipron, an oral glucagon like peptide-1 receptor agonist, is associated with improvements of CV risk biomarkers in participants with type 2 diabetes or obesity without diabetes. Cardiovasc Diabetol. 2025 Jun 6;24(1):240. doi: 10.1186/s12933-025-02781-x. PMID 40481478
- [Derived] Frias JP, Hsia S, Eyde S, Liu R, Ma X, Konig M, Kazda C, Mather KJ, Haupt A, Pratt E, Robins D. Efficacy and safety of oral orforglipron in patients with type 2 diabetes: a multicentre, randomised, dose-response, phase 2 study. Lancet. 2023 Aug 5;402(10400):472-483. doi: 10.1016/S0140-6736(23)01302-8. Epub 2023 Jun 24. PMID 37369232

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For maintenance doses of LY3502970: 3, 12, 24, 36, and 45 milligrams (mg), the initial dose will be 2 or 3 mg followed by additional escalation steps as appropriate. The dose escalation varied by dose group where the target maintenance dose was achieved between Weeks 4 and 12.
Groups:
- 3 mg LY3502970: Participants received maintenance dose of 3 mg with dose escalation starting from 2 mg LY3502970 administered orally once daily (QD).
Period: Overall Study
Arm/Group | Placebo | 3 mg LY3502970 | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 - 1 | 36 mg LY3502970 - 2 | 45 mg LY3502970 - 1 | 45 mg LY3502970 - 2 | 1.5 mg Dulaglutide
Started | 55 | 51 | 56 | 47 | 27 | 34 | 31 | 32 | 50
Received At Least One Dose of Study Drug | 55 | 51 | 56 | 47 | 27 | 34 | 31 | 32 | 50
Completed | 51 | 47 | 50 | 42 | 25 | 30 | 29 | 29 | 49
Not Completed | 4 | 4 | 6 | 5 | 2 | 4 | 2 | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 1 | 0 | 2 | 1 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Patient Decision due To Changes in Personal Life | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant was Unresponsive and Too Far Out of Window to Resume Treatment | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor decision due To inadvertent Enrollment | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant decided to Discontinue Treatment and only Return for Single Final Visit | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Site Terminated Participant due to Sponsor Directions | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- 3 mg LY3502970: Participants received maintenance dose of 3 mg with dose escalation starting from 2 mg LY3502970 administered orally QD.
- 1.5 mg Dulaglutide: Participants received 1.5 mg Dulaglutide administered SC QW.
- Total: Total of all reporting groups
Arm/Group | Placebo | 3 mg LY3502970 | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 - 1 | 36 mg LY3502970 - 2 | 45 mg LY3502970 - 1 | 45 mg LY3502970 - 2 | 1.5 mg Dulaglutide | Total
Number analyzed (Participants) | 55 | 51 | 56 | 47 | 27 | 34 | 31 | 32 | 50 | 383
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.30 (9.52) | 59.00 (9.43) | 57.40 (9.23) | 60.50 (9.11) | 59.20 (9.07) | 60.10 (9.37) | 58.10 (10.63) | 58.90 (8.18) | 58.80 (10.19) | 58.90 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 20 | 17 | 9 | 16 | 10 | 13 | 20 | 157
  Male | 28 | 26 | 36 | 30 | 18 | 18 | 21 | 19 | 30 | 226
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 7 | 15 | 5 | 6 | 7 | 7 | 6 | 7 | 74
  Not Hispanic or Latino | 41 | 44 | 41 | 42 | 21 | 27 | 24 | 26 | 43 | 309
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 4
  Asian | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 5 | 2 | 0 | 0 | 2 | 3 | 4 | 22
  White | 50 | 47 | 49 | 43 | 25 | 33 | 29 | 28 | 44 | 348
  More than one race | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 10 | 8 | 9 | 8 | 3 | 6 | 6 | 4 | 9 | 63
  Poland | 11 | 13 | 11 | 10 | 6 | 9 | 7 | 6 | 12 | 85
  Slovakia | 10 | 8 | 10 | 9 | 5 | 5 | 5 | 6 | 7 | 65
  United States | 24 | 22 | 26 | 20 | 13 | 14 | 13 | 16 | 22 | 170
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.1 (0.9) | 8.0 (0.8) | 8.2 (0.9) | 8.2 (0.9) | 8.0 (0.7) | 8.1 (0.8) | 8.3 (1.0) | 8.0 (0.8) | 8.0 (0.7) | 8.1 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c in LY3502970 as Compared to Placebo
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed model repeated measures (MMRM) model with Baseline + Country + Baseline HbA1c Group (<=8.0%, >8.0%) + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 26
Population: All participants who received at least one dose of LY3502970 or placebo and had baseline and at least one post-baseline value for HbA1c.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Groups:
- 3 mg LY3502970: Participants received maintenance dose of 3 mg with dose escalation starting from 2 mg LY3502970 administered orally once daily QD.
- 36 mg LY3502970: Participants received maintenance dose 36 mg with dose escalation starting from 2 mg, 3 mg, 6 mg, 8 mg, 12 mg, 24 mg and then 36 mg LY3502970 in LY 36mg-1 and dose escalation starting from 3 mg, 6 mg,12 mg, 24 mg and then 36 mg LY3502970 in LY 36mg-2 administered orally QD.
- 45 mg LY3502970: Participants received maintenance dose 45 mg with dose escalation starting from 3 mg, 6 mg, 8 mg, 12 mg, 24 mg, 36 mg and then 45 mg LY3502970 in LY 45mg-1 and dose escalation starting from 2 mg, 3 mg, 6 mg, 12 mg, 24 mg, 36 mg and then 45 mg LY3502970 in LY 45mg-2 administered orally QD.
Arm/Group | 3 mg LY3502970 | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 46 | 49 | 42 | 57 | 58 | 55
Percentage of HbA1c | -1.19 (0.137) | -1.91 (0.133) | -1.79 (0.149) | -2.03 (0.127) | -2.10 (0.124) | -0.43 (0.128)
Statistical Analysis 1: Comparison: 3 mg LY3502970 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.77, 95% CI 2-sided [-1.13 to -0.40]
Statistical Analysis 2: Comparison: 12 mg LY3502970 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.49, 95% CI 2-sided [-1.85 to -1.12]
Statistical Analysis 3: Comparison: 24 mg LY3502970 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.36, 95% CI 2-sided [-1.75 to -0.98]
Statistical Analysis 4: Comparison: 36 mg LY3502970 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.60, 95% CI 2-sided [-1.96 to -1.25]
Statistical Analysis 5: Comparison: 45 mg LY3502970 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.67, 95% CI 2-sided [-2.02 to -1.32]

2. Secondary Outcome: Change From Baseline in HbA1c in LY3502970 as Compared to Dulaglutide
Description: as for outcome 1
Time Frame: Baseline, Week 26
Population: All participants who received at least one dose of LY3502970 or dulaglutide, had a baseline, and at least one post-baseline value for HbA1c.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 3 mg LY3502970 | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | 1.5 mg Dulaglutide
Number analyzed (Participants) | 46 | 49 | 42 | 57 | 58 | 49
Percentage of HbA1c | -1.19 (0.137) | -1.91 (0.133) | -1.79 (0.149) | -2.03 (0.127) | -2.10 (0.124) | -1.10 (0.131)
Statistical Analysis 1: Comparison: 3 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Superiority; p = 0.626, Mixed Models Analysis; LS Mean Difference = -0.09, 95% CI 2-sided [-0.47 to 0.28]
Statistical Analysis 2: Comparison: 12 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.81, 95% CI 2-sided [-1.18 to -0.44]
Statistical Analysis 3: Comparison: 24 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.69, 95% CI 2-sided [-1.08 to -0.30]
Statistical Analysis 4: Comparison: 36 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.93, 95% CI 2-sided [-1.29 to -0.57]
Statistical Analysis 5: Comparison: 45 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.00, 95% CI 2-sided [-1.36 to -0.64]

3. Secondary Outcome: Percentage of Participants With HbA1c ≤ 6.5%
Description: Percentage of Participants with HbA1c ≤ 6.5%. Odds ratio was calculated using logistic regression model.
Time Frame: Week 26
Population: All participants who received at least one dose of study drug, had a baseline and at least one post-baseline HbA1c value.
Measure: Number; unit: Percentage of participants
Arm/Group | 3 mg LY3502970 | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo | 1.5 mg Dulaglutide
Number analyzed (Participants) | 46 | 49 | 42 | 57 | 58 | 22 | 49
Percentage of participants | 45.30 | 70.73 | 80.12 | 79.39 | 83.52 | 14.56 | 41.04
Statistical Analysis 1: Comparison: 3 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.77, 95% CI 2-sided [2.21 to 20.75]
Statistical Analysis 2: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 34.09, 95% CI 2-sided [9.92 to 117.16]
Statistical Analysis 3: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 48.33, 95% CI 2-sided [11.90 to 196.24]
Statistical Analysis 4: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 45.72, 95% CI 2-sided [13.61 to 153.64]
Statistical Analysis 5: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 77.23, 95% CI 2-sided [20.26 to 294.48]
Statistical Analysis 6: Comparison: 3 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p = 0.678, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.48 to 3.13]
Statistical Analysis 7: Comparison: 12 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.15, 95% CI 2-sided [2.19 to 17.24]
Statistical Analysis 8: Comparison: 24 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.71, 95% CI 2-sided [2.55 to 29.79]
Statistical Analysis 9: Comparison: 36 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.24, 95% CI 2-sided [3.05 to 22.30]
Statistical Analysis 10: Comparison: 45 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 13.93, 95% CI 2-sided [4.51 to 43.01]

4. Secondary Outcome: Percentage of Participants With HbA1c <7.0%
Description: Percentage of Participants with HbA1c <7.0%. Odds ratio was calculated using logistic regression model.
Time Frame: Week 26
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | 3 mg LY3502970 | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo | 1.5 mg Dulaglutide
Number analyzed (Participants) | 46 | 49 | 42 | 57 | 58 | 55 | 49
Percentage of participants | 65.17 | 78.92 | 91.24 | 92.75 | 95.76 | 24.27 | 64.06
Statistical Analysis 1: Comparison: 3 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.19, 95% CI 2-sided [2.93 to 22.90]
Statistical Analysis 2: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 25.02, 95% CI 2-sided [7.57 to 82.69]
Statistical Analysis 3: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 62.31, 95% CI 2-sided [12.26 to 316.63]
Statistical Analysis 4: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 67.57, 95% CI 2-sided [17.56 to 259.97]
Statistical Analysis 5: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 129.55, 95% CI 2-sided [26.72 to 628.09]
Statistical Analysis 6: Comparison: 3 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p = 0.802, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.43 to 2.96]
Statistical Analysis 7: Comparison: 12 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p = 0.026, Regression, Logistic; Odds Ratio (OR) = 3.46, 95% CI 2-sided [1.16 to 10.31]
Statistical Analysis 8: Comparison: 24 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 8.61, 95% CI 2-sided [1.83 to 40.51]
Statistical Analysis 9: Comparison: 36 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 9.34, 95% CI 2-sided [2.67 to 32.71]
Statistical Analysis 10: Comparison: 45 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 17.90, 95% CI 2-sided [4.02 to 79.70]

5. Secondary Outcome: Change From Baseline in Fasting Serum Glucose
Description: Fasting glucose is a test to determine sugar levels in blood sample after an overnight fast. LS mean was determined by MMRM model with Baseline + Country + Baseline HbA1c Group (<=8.0%, 8.0%) + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 26
Population: All participants who received at least one dose of study drug, had baseline and at least one post-baseline fasting glucose data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 3 mg LY3502970 | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo | 1.5 mg Dulaglutide
Number analyzed (Participants) | 46 | 49 | 42 | 57 | 58 | 55 | 49
milligrams per deciliter (mg/dL) | -32.6 (4.14) | -53.7 (3.92) | -52.2 (4.49) | -53.9 (3.79) | -55.9 (3.69) | -11.1 (3.90) | -33.2 (3.91)
Statistical Analysis 1: Comparison: 3 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -21.5, 95% CI 2-sided [-32.7 to -10.3]
Statistical Analysis 2: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -42.5, 95% CI 2-sided [-53.4 to -31.7]
Statistical Analysis 3: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -41.0, 95% CI 2-sided [-52.7 to -29.3]
Statistical Analysis 4: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -42.7, 95% CI 2-sided [-53.5 to -32.0]
Statistical Analysis 5: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -44.7, 95% CI 2-sided [-55.3 to -34.2]
Statistical Analysis 6: Comparison: 3 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = 0.6, 95% CI 2-sided [-10.6 to 11.8]
Statistical Analysis 7: Comparison: 12 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -20.5, 95% CI 2-sided [-31.4 to -9.5]
Statistical Analysis 8: Comparison: 24 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p = 0.002, Mixed Models Analysis; LS Mean Difference = -19.0, 95% CI 2-sided [-30.7 to -7.2]
Statistical Analysis 9: Comparison: 36 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -20.7, 95% CI 2-sided [-31.4 to -9.9]
Statistical Analysis 10: Comparison: 45 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -22.7, 95% CI 2-sided [-33.2 to -12.1]

6. Secondary Outcome: Change From Baseline in Body Weight
Description: LS mean was determined by MMRM model with Baseline + Country + Baseline HbA1c Group (<=8.0%, >8.0%) + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 26
Population: All participants who received at least one dose of study drug, had baseline and at least one post-baseline body weight data.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 3 mg LY3502970 | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo | 1.5 mg Dulaglutide
Number analyzed (Participants) | 50 | 53 | 46 | 57 | 62 | 55 | 50
kilograms (kg) | -3.7 (0.79) | -6.5 (0.76) | -9.7 (0.85) | -9.5 (0.73) | -10.1 (0.71) | -2.2 (0.74) | -3.9 (0.76)
Statistical Analysis 1: Comparison: 3 mg LY3502970 vs Placebo; Test type: Other; p = 0.153, Mixed Models Analysis; LS Mean Difference = -1.6, 95% CI 2-sided [-3.7 to 0.6]
Statistical Analysis 2: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -4.3, 95% CI 2-sided [-6.4 to -2.2]
Statistical Analysis 3: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -7.6, 95% CI 2-sided [-9.8 to -5.3]
Statistical Analysis 4: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -7.4, 95% CI 2-sided [-9.4 to -5.3]
Statistical Analysis 5: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -7.9, 95% CI 2-sided [-9.9 to -5.9]
Statistical Analysis 6: Comparison: 3 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p = 0.914, Mixed Models Analysis; LS Mean Difference = 0.1, 95% CI 2-sided [-2.0 to 2.3]
Statistical Analysis 7: Comparison: 12 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p = 0.015, Mixed Models Analysis; LS Mean Difference = -2.6, 95% CI 2-sided [-4.7 to -0.5]
Statistical Analysis 8: Comparison: 24 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -5.9, 95% CI 2-sided [-8.1 to -3.6]
Statistical Analysis 9: Comparison: 36 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -5.7, 95% CI 2-sided [-7.8 to -3.6]
Statistical Analysis 10: Comparison: 45 mg LY3502970 vs 1.5 mg Dulaglutide; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -6.2, 95% CI 2-sided [-8.3 to -4.2]

7. Secondary Outcome: Pharmacokinetics (PK): Steady State Area Under the Concentration Curve (AUC) of LY3502970
Description: PK: Steady State AUC of LY3502970
Time Frame: Pre-dose (Week (wk) 0, wk 8, wk 12, and wk 26); Post-dose (wk 4, wk 8, wk 16, wk 20, and end of treatment).
Population: All participants who received at least one dose of LY3502970 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram *hour per milliliter (ng*h/mL)
Arm/Group | 3 mg LY3502970 | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 - 1 | 36 mg LY3502970 - 2 | 45 mg LY3502970 - 1 | 45 mg LY3502970 - 2
Number analyzed (Participants) | 45 | 48 | 43 | 24 | 29 | 25 | 28
nanogram *hour per milliliter (ng*h/mL) | 364 (38.7) | 1020 (63.5) | 1500 (84.5) | 1830 (94.6) | 2430 (39.8) | 2230 (80.4) | 2550 (55.3)

ADVERSE EVENTS:
Time Frame: Baseline Through Safety Follow-Up (Up To Week 28)
Description: All randomized participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Placebo | 3 mg LY3502970 | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 - 1 | 36 mg LY3502970 - 2 | 45 mg LY3502970 - 1 | 45 mg LY3502970 - 2 | 1.5 mg Dulaglutide
All-Cause Mortality (participants affected / at risk) | 1/55 | 0/51 | 0/56 | 0/47 | 0/27 | 0/34 | 0/31 | 0/32 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/55 | 3/51 | 1/56 | 5/47 | 1/27 | 1/34 | 0/31 | 1/32 | 1/50
Other Adverse Events (participants affected / at risk) | 25/55 | 34/51 | 40/56 | 32/47 | 21/27 | 18/34 | 21/31 | 23/32 | 23/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=55) | 3 mg LY3502970 (N=51) | 12 mg LY3502970 (N=56) | 24 mg LY3502970 (N=47) | 36 mg LY3502970 - 1 (N=27) | 36 mg LY3502970 - 2 (N=34) | 45 mg LY3502970 - 1 (N=31) | 45 mg LY3502970 - 2 (N=32) | 1.5 mg Dulaglutide (N=50)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pylorospasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=55) | 3 mg LY3502970 (N=51) | 12 mg LY3502970 (N=56) | 24 mg LY3502970 (N=47) | 36 mg LY3502970 - 1 (N=27) | 36 mg LY3502970 - 2 (N=34) | 45 mg LY3502970 - 1 (N=31) | 45 mg LY3502970 - 2 (N=32) | 1.5 mg Dulaglutide (N=50)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (5) | 1 (2) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 7 (9) | 7 (8) | 6 (7) | 6 (6) | 1 (1) | 1 (1) | 4 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 11 (18) | 9 (10) | 7 (11) | 7 (8) | 2 (3) | 9 (10) | 9 (11) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 6 (6) | 4 (4) | 3 (3) | 3 (5) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (3) | 3 (3) | 5 (11) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 4 (5) | 3 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (4) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 12 (15) | 21 (27) | 16 (20) | 10 (20) | 9 (18) | 9 (15) | 8 (9) | 9 (13)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 12 (16) | 13 (16) | 9 (28) | 7 (9) | 11 (18) | 7 (10) | 4 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3) | 5 (5) | 0 (0) | 1 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0/27 (0) | 0/25 (0) | 0/20 (0) | 0/17 (0) | 0/9 (0) | 0/16 (0) | 0/10 (0) | 0/13 (0) | 1/20 (1)
Covid-19 (Infections and infestations) | 3 (3) | 2 (2) | 5 (5) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 2 (2) | 5 (5) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (4) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 3 (4) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 7 (9) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 0/28 (0) | 0/26 (0) | 0/36 (0) | 0/30 (0) | 0/18 (0) | 1/18 (1) | 0/21 (0) | 0/19 (0) | 0/30 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT05048719/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT05048719/SAP_001.pdf